CLINICAL TRIAL: NCT05778968
Title: The Effect of Different Etco2 Levels on the End-tidal Concentration of Sevoflurane in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Etco2 Levels on the End-tidal Concentration of Sevoflurane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MAC of sevoflurane
Record Dates: First submitted 2023-03-08; First posted 2023-03-22 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: End-tidal Sevoflurane; End-tidal Carbon Dioxide; Minimum Alveolar Concentration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low ETCO2 (Active Comparator)
  Interventions: Procedure: low etco2
- normal ETCO2 (Active Comparator)
  Interventions: Procedure: normal etco2
- high ETCO2 (Active Comparator)
  Interventions: Procedure: high etco2

INTERVENTIONS:
Procedure: low etco2 — Etco2 levels will be adjusted at levels ranging between 25 mm Hg and 30 mm Hg
  Arms: low ETCO2
Procedure: normal etco2 — Etco2 levels will be adjusted at levels ranging between 31 mm Hg and 40 mm Hg
  Arms: normal ETCO2
Procedure: high etco2 — Etco2 levels will be adjusted at levels ranging between 41 mm Hg and 45 mm Hg
  Arms: high ETCO2

SUMMARY:
he assessment of adequate levels of anaesthesia traditionally relies not only on a patient's movement but also on the hemodynamic response (or both) to a surgical stimulus

DETAILED DESCRIPTION:
Currently a derivative of MAC namely, end tidal partial pressure (FET) displayed on the work station as concentration , maybe an alternative useful measure of the anaesthetic effect of an inhaled anaesthetic agent

. Many pharmacological factors have been associated with alterations in MAC and Mac derivatives such as nonsteroidal anti-inflammatory drugs (NSAIDs), analgesics, and anesthetics.

However, few studies have focused on physiological factors, such as hypercarbia or hypocarbia. A correlation has been found between Paco2 and Etco2 in ventilated patients with healthy lungs. Some authors have suggested that Etco2 could be considered appropriate for estimating Paco2 even in critical patients. Knowledge of the effects of Paco2 on end tidal concentration of sevoflurane among patients undergoing laparoscopic cholecystectomy may help anaesthesiologists titrate sevoflurane carefully and precisely during different mechanical ventilation settings to avoid dose-dependent hypotension, impaired cardiac contractility, and hypothermia caused by excessive anaesthetic depth of sevoflurane.

ELIGIBILITY:
Inclusion Criteria:

* American Society of anaesthesiologist ASA physical status I, II
* admitted for laparoscopic cholecystectomy

Exclusion Criteria:

* Refusal of patients.

  * Patients with renal or liver dysfunction.
  * Patients with chronic pain other than cholelithiasis.
  * Cardiac disorders as uncontrolled hypertension, arrhythmia, Ischaemic heart disease, valvular heart disease and pulmonary hypertension.
  * Patient with haematological disorder as Sickle cell disease.
  * Chest patient as asthma, COPD.
  * Combined surgery .
  * History of allergy to any of the study drugs.
  * Patients with communication problems, cognitive dysfunction, or psychological disorders.
  * Patients who received analgesics or sedatives 24 h before a scheduled surgery.
  * Alcohol or drug abuse.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
end tidal concentration of sevoflurane | Total time of operation
  end tidal concentration of sevoflurane is measured by multiple gas analyser during operation

CONTACTS AND LOCATIONS:
Overall Officials: thanaa elnomany, MD, Study Director — tanta university, faculty of medicine
Locations (1):
- tarek Abdelhay Mostafa, Tanta, El Gharbyia, Egypt

IPD SHARING:
Plan to Share IPD: No